CLINICAL TRIAL: NCT00102583
Title: A Phase I Clinical Trial to Study the Safety of a Sustained-Release Subconjunctival Cyclosporine Implant for Ocular Graft-vs-Host Disease (GVHD1)
Brief Title: Cyclosporine Implant for Ocular Graft-Versus-Host Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 050002; 05-EI-0002
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-03-15

CONDITIONS: Graft Vs Host Disease
Keywords: Dry Eye; Lacrimal Gland; Tear Deficiency; Keratitis Sicca; GVHD; Ocular GVHD; Ocular Graft Vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease; Dry Eye Syndromes; Keratitis sicca

INTERVENTIONS:
Drug: Subconjunctival Cyclosporine Implant

SUMMARY:
Graft-vs.-Host Disease (GVHD) is a major complication of allogeneic hematopoietic stem cell transplantation (SCT) commonly affecting the skin, liver, gastrointestinal tract, and eye. The most common clinical manifestations of ocular GVHD generally result from

involvement of the lacrimal gland and the conjunctiva. Lacrimal gland involvement can lead to aqueous tear deficiency resulting in severe keratoconjunctivitis sicca (KCS) which can significantly increase the morbidity of patients with chronic GVHD.

Systemic immunosuppressants such as cyclosporine (CsA) can be effective for treating ocular GVHD including lacrimal gland dysfunction. However, systemic immunosuppression is not generally prescribed for patients whose sole manifestation of GVHD is ocular complications as it may negate the overall graft-vs.-tumor effect and decrease patient survival. Topical CsA and corticosteroids are generally not effective for treating aqueous tear deficiency possible due to epithelial barriers preventing penetration of the drugs to the lacrimal gland. A sustained-release subconjunctival CsA implant was developed to bypass these epithelial barriers and significantly increase the CsA concentrations in the lacrimal gland to treat aqueous tear deficiency related to GVHD.

The objective of this randomized pilot study is to investigate the safety and potential efficacy of a CsA implant in patients with lacrimal gland involvement and aqueous tear deficiency related to GVHD. Safety will be evaluated in terms of adverse events related to the implant. Efficacy will be evaluated by changes in Schirmer tear test (with anesthesia). Secondary efficacy evaluation will include changes in corneal and conjunctival staining grades, best-corrected visual acuity (BCVA), the Ocular Surface Disease Index (OSDI), changes in conjunctival GVHD grades, tear break-up time and meibomian gland dysfunction.

Patients with active systemic GVHD with aqueous tear deficiency associated with lacrimal gland dysfunction following allogeneic hematopoietic SCT who are nine years of age or older are eligible for inclusion in this pilot study. The study will involve surgical placement of the CsA implant into the subconjunctival space adjacent to the lacrimal gland of one eye in each participant. Participants older than 12 years of age will be randomized to receive one of two implant release rates. All participants under the age of 12 will receive the smaller, lower dose implant. However, all participants under age 12 will not be randomized and will only be eligible to receive the smaller, lower dose implant.

The implant will remain in place for up to two years and then be removed. IF the participant has clinical success, they will be given the option of allowing the implant to remain in place for an additional year. Clinical success is achieved if the participant meets any of the following measures in either eye assessed at the 1-year visit:

Interval change from baseline characteristics

Decrease in corneal staining by greater than or equal to 2

Decrease in temporal or nasal conjunctival staining grades by greater than or equal to 2

Decrease in total staining grade by greater than or equal to 2

Decrease in OSDI calculated score by greater than or equal to 20%

Increase in Schirmer tear test measurement by greater than or equal to 3 mm

Meets mild-moderate KCS characteristics at 1 year

Corneal staining grade less than or equal to 3

Nasal or temporal conjunctival staining grades less than or equal to 3

OSDI calculated score less than or equal to 15

Schirmer tear test measurement greater than or equal to 5 mm

For participants with implant duration of one year, safety evaluations will be conducted at baseline (pre-implantation) and monthly post-implantation for 13 months. Additional safety assessments will be done at 1 day, and at 1 and 2 weeks post-operatively for implant placement and removal procedures. Safety and efficacy evaluations will be conducted at baseline, at 1, 3, 6, 9, and 12 months post-implantation, and at 3 months following implant removal (15 months post-implantation). For participants with clinical success and who choose the implant to remain for another year, visits will be held as described above then conducted at 2-month intervals starting at month 14. Safety evaluations will be conducted every 2 months until the end of the second year. Additional safety assessments will be done at 1 day, and at 1 and 2 weeks post-operatively for implant removal procedures. Safety and efficacy evaluations will be conducted at 16, 20, and 24 months post-implantation, and at 3 months following implant removal (27 months post-implantation).

DETAILED DESCRIPTION:
The objective of this randomized pilot study is to investigate the safety and potential efficacy of a CsA implant in participants with lacrimal gland involvement and aqueous tear deficiency related to GVHD. Safety will be evaluated in terms of adverse events related to the implant. Efficacy will be evaluated by changes in Schirmer tear test (with anesthesia). Secondary efficacy evaluation will include changes in corneal and conjunctival staining grades, best-corrected visual acuity (BCVA), the Ocular Surface Diseases Index (OSDI), changes in conjunctival GVHD grades, tear break-up time and meibomian gland dysfunction.

Participants with active systemic GVHD with aqueous tear deficiency associated with lacrimal gland dysfunction following allogeneic hematopoietic SCT who are nine years of age or older are eligible for inclusion in this pilot study. The study will involve surgical placement of the CsA implant into the subconjunctival space adjacent to the lacrimal gland of one eye in each participant. Participants older than 12 years of age will be randomized to receive one of two implant release rates. However, all participants under age 12 will not be randomized and will only be eligible to receive the smaller, lower dose implant. On each anniversary study visit a participant will be given the opportunity to retain the implant on an annual basis. This will be based upon the determination of clinical success (defined in the Study Design section below) combined with a participant's report of symptom improvement. The Implant will be removed if the Investigator believes the implant is harmful or if the participant requests the implant to be removed.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for the study each participant must satisfy all of the following inclusion criteria:

* Male or female greater than or equal to 9 years of age.
* Must be greater than or equal to 30 days post-hematopoietic stem cell transplantation (SCT) and have systemic GVHD diagnosed by the transplant physician.
* Must have lacrimal gland dysfunction from GVHD following SCT as defined by Schirmer tear test score (with anesthesia) of greater than or equal to 1 mm but less than or equal to 9 mm in both eyes.
* Must have open puncta and no puncta plug placement at the time of enrollment.
* If using topical corticosteroids, must be equal dose in both eyes of less than or equal to 4 drops per day.
* Topical lubrication using tear substitutes (includes eye drops, gels, and ointments) are permitted with equal dosing in both eyes.
* Must understand and sign informed consent or assent.
* Must be willing and able to comply with study evaluation and testing schedule.
* Females of childbearing potential and all males must agree to use an effective form of birth control for duration of the study.
* Females of childbearing potential must have a negative serum pregnancy test at baseline evaluation.

EXCLUSION CRITERIA:

To be eligible for the study, participants must not satisfy any of the following exclusion criteria.

* Use of a topical ophthalmic cyclosporine formulation less than or equal to 30 days prior to enrollment.
* Diagnosed with active ocular infection.
* History of recurrent herpes keratitis or active disease less than or equal to 6 months prior to enrollment.
* Aqueous tear deficiency or KCS related to previous irradiation, Stevens-Johnson syndrome, cicatricial pemphigoid, alkali burns, trachoma or Sjogren's syndrome.
* Seropositive for Hepatitis C (i.e. positive anti-HCV antibody) or seropositive for HIV with testing performed no earlier than 4 months before the date of stem cell transplantation.
* Diagnosis of active sarcoidosis.
* Use of a drug with anticholinergic activity within less than 4 times the half-life of the drug prior to enrollment (e.g., carbamazepine [Tegretol (R)] has a half-life of 16-24 hours so must not be used within 4 days of enrollment).
* Use of an investigational drug for eye disease within 30 days of enrollment.
* Known allergy or hypersensitivity to cyclosporine, fluorescein, or lissamine green.
* Uncontrolled systemic disease or serious illness that could, in the investigator's opinion, interfere with the participant's ability to comply with study therapy, required follow-up testing, or interfere with interpretation of the study results.
* Pregnant or lactating female.
* Serum creatinine greater than 2.5 mg/dL, absolute neutrophil count (ANC) less than 750/MicroL Platelet count less than 25,000/MicroL, Partial Thromboplastin Time (PTT), or International Normal Ratio (INR) or Prothrombin Time (PT) exceeding the institutional upper limit of normal would require review by the Hematologist for surgical clearance. Hematologist review of the abnormal coagulation value and approval for surgery must be documented in the medical record prior to the surgical procedure.
* Participants that have received total body irradiation or direct eye/orbital radiation greater than 5000 cGy. (Potential participants will be assessed by a study clinician to determine that the cause of the dry eye symptoms is due to GVHD and not radiation. The clinician, in conjunction with the oncology staff as needed, will also assess the participant's clinical exam and medical history).

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2004-10-14; Primary Completion 2011-03-15 (Actual); Study Completion 2011-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bhushan V, Collins RH Jr. Chronic graft-vs-host disease. JAMA. 2003 Nov 19;290(19):2599-603. doi: 10.1001/jama.290.19.2599. No abstract available. PMID 14625337
- [Background] Ogawa Y, Okamoto S, Wakui M, Watanabe R, Yamada M, Yoshino M, Ono M, Yang HY, Mashima Y, Oguchi Y, Ikeda Y, Tsubota K. Dry eye after haematopoietic stem cell transplantation. Br J Ophthalmol. 1999 Oct;83(10):1125-30. doi: 10.1136/bjo.83.10.1125. PMID 10502571
- [Background] Young NS, Barrett AJ. The treatment of severe acquired aplastic anemia. Blood. 1995 Jun 15;85(12):3367-77. No abstract available. PMID 7780125